CLINICAL TRIAL: NCT04019574
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Four-way Crossover Study to Investigate the Effects of Single Intravenous Doses of Difelikefalin (CR845) on the QTc Interval in Healthy Subjects
Brief Title: Study to Investigate the Effects of Single Intravenous Doses of Difelikefalin (CR845) on the QTc Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR845-100201
Record Dates: First submitted 2019-07-08; First posted 2019-07-15 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Difelikefalin; CR845; QTc; TQT
MeSH Terms: interventions — difelikefalin; Moxifloxacin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CR845 0.5 mcg/kg IV (Therapeutic Dose) (Experimental)
  Interventions: Drug: CR845 0.5 mcg/kg IV
- CR845 3 mcg/kg IV (Supratherapeutic Dose) (Experimental)
  Interventions: Drug: CR845 3 mcg/kg IV
- Placebo IV (Placebo Comparator)
  Interventions: Other: Placebo
- Moxifloxacin 400 mg (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg Oral Tablet

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg IV — 0.5 mcg/kg IV CR845
  Other Names: Difelikefalin 0.5 mcg/kg
  Arms: CR845 0.5 mcg/kg IV (Therapeutic Dose)
Drug: CR845 3 mcg/kg IV — 3 mcg/kg IV CR845
  Other Names: Difelikefalin 3 mcg/kg
  Arms: CR845 3 mcg/kg IV (Supratherapeutic Dose)
Drug: Moxifloxacin 400 mg Oral Tablet — 400 mg Oral Moxifloxacin
  Other Names: Avelox
  Arms: Moxifloxacin 400 mg
Other: Placebo — IV Placebo as a bolus injection
  Arms: Placebo IV

SUMMARY:
This is a Phase 1, randomized, double-blind (except for moxifloxacin), placebo- and positive-controlled, single-site, 4-way crossover study to investigate the effects of single therapeutic and supratherapeutic IV doses of difelikefalin (CR845) on the QTc interval in healthy adult subjects. Subjects will be randomized to a treatment sequence consisting of 4 treatment periods with a minimum 5-day washout between treatments. Subjects will receive each of the study treatments over the course of the study. Randomized subjects will receive the assigned study treatment as a single dose in the fasted state in the morning on Day 1 of each treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight between 50 to 120 kg and body mass index within 18 to 29 kg/m2 at Screening;
* Current nonsmokers who have not used any tobacco- or nicotine-containing products (chewed or smoked) or replacement products, including, but not limited to, electronic cigarettes, in the 45 days prior to Screening.

Key Exclusion Criteria:

* Past or present diseases, which as judged by the Investigator, may affect the outcome of this study;
* Any condition or situation that, in the opinion of the Investigator, would prevent proper evaluation of the safety or efficacy of the study treatment according to the study protocol;
* History of hypersensitivity or allergy to moxifloxacin or any other study treatment or history of tendonitis or tendon rupture with moxifloxacin or any other quinolone type drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
QTc change from baseline following CR845 treatment. | Baseline, Day 1

SECONDARY OUTCOMES:
Change from baseline in QTc with Bazett correction (QTcB). | Baseline, Day 1
Change from baseline in Heart Rate. | Baseline, Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (1):
- Cara Therapeutics Study Site, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No